CLINICAL TRIAL: NCT02288299
Title: Long-Term Effect of LIAM (Lung Insufflation Assist Maneuver) on Respiratory Performance in Non-invasive Ventilated Patients Suffering From Neuromuscular Disease
Brief Title: Long-Term Effect of LIAM on Respiratory Performance in NIV Patients Suffering From Neuromuscular Disease
Acronym: LIAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01005-42
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-02

CONDITIONS: Neuromuscular Disease
Keywords: Instrumental cough assistance; positive pressure insufflation maneuver; home mechanical ventilation; prospective evaluation
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- non invasive mechanical ventilation (Experimental): Patients suffering from neuromuscular disease with NIV indication and cough inefficiency
  Interventions: Device: non invasive mechanical ventilation

INTERVENTIONS:
Device: non invasive mechanical ventilation — instrumental increase of inspiratory capacity and cough

SUMMARY:
The long-term effect of LIAM (Lung Insufflation Assist Maneuver) on respiratory performance in home non-invasively ventilated (NIV) patients suffering from neuromuscular disease will be assessed in a prospective, randomized, cross over, open label study

DETAILED DESCRIPTION:
In advanced neuromuscular disorders, respiratory complications represent the main cause of morbidity and mortality. Beside chronic respiratory insufficiency, necessitating a ventilatory support, mostly performed by non-invasive ventilation (NIV), cough is impaired due to the muscle weakness, and respiratory physiotherapy becomes an essential part of the management.

Various techniques have been proposed to improve lung recruitment and cough in neuromuscular patients. The assisted techniques based on a positive pressure insufflation maneuver have shown an improvement in physiological variables on the short term, but there is to date no good-quality prospective study allowing to evaluate the long term efficacy of mechanical cough assistance devices in neuromuscular patients.

We designed a randomized, cross over, open label study to assess the long-term effect of LIAM (Lung Insufflation Assist Maneuver) on respiratory performance in NIV patients suffering from neuromuscular disease.

ELIGIBILITY:
Inclusion Criteria:

* o neuromuscular disease ( progressive muscular dystrophy, for example; Duchenne muscular dystrophy, spinal muscular atrophy)

  * age ≥ 18 years
  * indication to NIV (ongoing ventilation or new patients)
  * vital capacity ≤ 50% pred
  * peak cough flow < 270 l/min
  * "LIAM Responder" = increased insufflation capacity (≥ + 50%) and Peak Cough Flow (PCF ≥+ 50%) with LIAM

Exclusion Criteria:

* o acute respiratory failure (respiratory acidosis)

  * home treatment by instrumental cough assistance in the preceding 12 months
  * ongoing medical treatment of the neuromuscular disease (for ex: corticosteroids in Duchenne disease, enzyme therapy in Pompe disease)
  * previous pneumothorax
  * plan of legal protection
  * pregnant or breastfeeding women
  * failure to cooperate
  * no affiliation to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10-29 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the maximal assisted vital capacity (maximal insufflation capacity) between the begin of the treatment period and the 3-months follow up | 15 minutes
  Change in the maximal assisted vital capacity (maximal insufflation capacity) between the begin of the treatment period and the 3-months follow up

SECONDARY OUTCOMES:
spontaneous vital capacity | 15 minutes
  spontaneous vital capacity change at 3 months
peak flow | 15 minutes
  peak cough flow (spontaneous / assisted) change at 3 months
optoelectronic plethysmography | 1 hour
  change at 3 months in the distribution in ventilation (assessed by optoelectronic plethysmography), spontaneous/assisted

CONTACTS AND LOCATIONS:
Overall Officials: David Orlikowski, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Home ventilation Unit , Raymond Poincaré hospital, Garches, Paris Area, France